CLINICAL TRIAL: NCT06959680
Title: The Effect of Kinesiotaping on Posture and Balance in Patients With Postural Thoracic Hyperkyphosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Feyza Nur Yucel, Principal Investigator, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2024.256
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Kyphosis Thoracic; Kyphosis Postural Thoracic; Kinesio Taping; Postural Kyphosis; Balance
Keywords: Balance; Postural Kyphosis; Kinesio taping
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: There are 3 groups of participants in the study Group 1 participants will receive exercise therapy alone. Group 2 participants will receive exercise and kinesiotaping treatment. Group 3 participants will receive exercise and shamtaping treatment.
Who Masked: Participant, Care Provider
Masking Description: Controlled Randomized Single-Blind Prospective Cohort One group does not know whether the other group received taping treatment. The physiotherapist also does not know whether a participant received taping therapy.
  The physiotherapist only teaches the participants exercises
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 Exercise (Active Comparator): Group 1 participants will receive exercise therapy alone.
  Interventions: Other: Exercise
- Group 2 Exercise and Kinesiotaping (Active Comparator): Group 2 participants will receive exercise and kinesiotaping treatment.
  Interventions: Other: Exercise and Kinesiotaping
- Group 3 Exercise and Shamtaping (Sham Comparator): Group 3 participants will receive exercise and shamtaping treatment.
  Interventions: Other: exercise and sham taping

INTERVENTIONS:
Other: Exercise and Kinesiotaping — Exercise and Kinesiotaping
  Arms: Group 2 Exercise and Kinesiotaping
Other: Exercise — only exercise will be performed without any band treatment
  Arms: Group 1 Exercise
Other: exercise and sham taping — exercise and sham banding (banding without tension with plaster)
  Arms: Group 3 Exercise and Shamtaping

SUMMARY:
The primary aim of our research is to evaluate the positive effects of exercise and kinesiotaping on the thoracic kyphosis angle in young adults between the ages of 18-45 with a thoracic kyphosis angle of 40 degrees and above. Secondary aims are to investigate the effects of kinesiotaping on dynamic and static balance, pain, and quality of life in patients with thoracic hyperkyphosis.

DETAILED DESCRIPTION:
In young adults, the thoracic kyphosis angle varies between 20-45◦ and 40◦ and above is defined as thoracic hyperkyphosis. The prevalence of thoracic hyperkyphosis is between 20-40% and is most commonly idiopathic . Thoracic hyperkyphosis is associated with back pain, limitation of movement-function, loss of balance, decreased quality of life and increased risk of falls. In the absence of pain or loss of function, especially young patients may present to improve cosmetic appearance. In the first stage of treatment, exercise, manual therapy, and in advanced stages, bracing and surgery can be applied . In treatment to reduce kyphosis, exercise is recommended at all ages and bracing is recommended in selected patients who do not respond to exercise. Multimodal combination therapies have been shown to be effective in young people . Kinesiobanding (KT) is an application that supports fascia, muscles and joints and reduces pain and inflammation . The combination of taping and exercise has been shown to have a positive effect on balance in hyperkyphotic adolescents. There is no study in the literature evaluating the effects of kinesiobanding on both balance parameters and kyphosis angle in young adults with thoracic hyperkyphosis. We think that favorable results can be obtained in the young age group with this study and our study may provide findings that kinesiobanting can be added to exercise therapy in routine treatment.

Sample Size of the Study: The sample size was determined by G-power analysis using the reference article. The number of participants to be included in the study was calculated as 16 patients for each group with G-power with a power of 95% and a type 1 error of 0.05 .

Patients will be divided into 3 groups. Taking into account the 20% loss rate that may occur during follow-up, a total of 48 patients were planned to be included in the study for 3 groups; 16 patients in each group.

TREATMENT GROUPS:

Group 1 (n=16)(E): exercise Group 2 (n=16)(E+KT): exercise + kinesio taping Group 3 (n=16)(E+SH): exercise + sham taping

The study groups will be determined according to the eligibility criteria among patients who present to the Physical Medicine and Rehabilitation outpatient clinic with complaints of posture disorder or nonspecific back pain and who have a thoracic kyphosis angle of 40 degrees or more on lateral radiography.

Cobb Angle Measurement:

Thoracic kyphosis angle will be measured on thoracic lateral radiograph. According to the literature, the gold standard measurement method is Cobb angle measurement; since the T4-T12 vertebra angle is less visible above the T4 vertebra level due to the superposition of other structures, the T4-T12 vertebra angle is used. The angle at the intersection point of the lines drawn parallel to the upper endplate of the T4 vertebra and the lower endplate of the T12 vertebra gives the Cobb angle . Patients with a Cobb angle of 40 and above and who do not have any additional disease to explain pain or hyperkyphosis will be included in the study.

Grouping of Participants, Patient Follow-up Form and Evaluations Our study was planned as a randomized single-blind prospective cohort, double-center study. Between 23/11/2024 - 23/08/2025 patients who meet the inclusion criteria among young adults aged 18-45 years who applied to Marmara University Faculty of Medicine and Sultan Abdulhamid Han Training and Research Hospital Physical Medicine and Rehabilitation outpatient clinics with complaints of nonspecific back pain or posture disorder will be included in the study. The study is planned to last 9 months.

Cobb angle measurement on thoracic lateral radiograph, kyphosis angle and index measurement with Flexicurve device, Biodex device, VAS scoring, Berg balance scale, SRS-22 questionnaire, International Physical Activity Questionnaire (Short) (IPAQ) will be used in the study.

Informed consent: After the patients are verbally informed, consent forms will be given to the patients in which the purpose of the study is clearly explained and they will be asked to sign the forms.

Exercise Program (1st group=E group) The exercises were designed as a 4-week home program. In all three groups, the exercises will be performed once a day, 3 days a week, one day apart, for 4 weeks.

Each exercise will be performed with 10 repetitions in the first two weeks and 15 repetitions in the third and fourth weeks, with 5 sec contraction and 5 sec relaxation, with a 1 min break between two different exercises.

In the first stage, home exercises will be demonstrated to the patients. Afterwards, all patients will be given a pictorial exercise brochure and an exercise diary; patients will be encouraged to comply with the treatment with weekly phone calls.

In postural thoracic hyperkyphosis, strengthening, stretching exercises and breathing exercises will be given for the most affected muscle groups. Posture exercises were planned for trapezius, lattismus dorsi, levator scapula, rhomboids, serratus posterior-superior-inferior, longissimus thoracis, spinalis thoracis, iliocostalis thoracis, semispinalis thoracis, multifidus, rotatores thoracis, diaphragm, intercostal externi, abdominal muscles:

* Thoracic and shoulder girdle strengthening exercises
* Pelvic and lumbar stabilization exercises
* Anterior and lateral abdominal muscle strengthening exercises
* Hip flexor stretching exercises
* Lumbar extensor stretching exercises
* Breathing exercises Kinesio Taping (2nd Group= E+KT Group) Kinesiobant will first be tested on a small area of the forearm and treatment will be discontinued if allergy develops. Taping will be applied with the patient in upright posture and shoulders in retraction. From the level of the acromioclavicular joint, the first 5 cm will be applied without stretching, then maximum stretching will be applied, moving to the diagonal and ending at the lower border of the costa, the adhesion point will be adhered without stretching. The same process will be applied on the opposite side and a total of two I-shaped bands will be used to create an X-shape on the back. The crossing point of the bands will be adjusted to the lower 1/3 of the medial edge of the scapula. Taping will be performed after all initial measurements (T0) and will be renewed weekly (on days 0, 7, 14, 21). At the end of the 1st month, i.e. on day 28 (T1), the last measurements will be made with the kinesio tape and then the tape will be removed. One month after the end of the treatment, the patient will be called again (T2) and final measurements will be made without the tape.

Sham Taping (3rd group= E+SH group) Sham taping treatment will be performed to exclude the biofeedback effect of taping and to distinguish its functional effect. The patch to be used in sham taping will first be tested on a small area of the forearm and if allergy develops, the treatment will be terminated. Taping will be applied with the patient in upright posture and shoulders in retraction. Skin color, elasticity and non-stretchable plaster of the same color as the skin will be used. From the level of the acromioclavicular joint, it will be applied from the level of the acromioclavicular joint to the diagonal without stretching and will be adhered to the adhesion point without stretching, ending at the lower border of the costa. The same procedure will be applied to the opposite side and an X shape will be formed on the back using a total of two I-shaped plasters. The crossing point of the bands will be adjusted to the lower 1/3 of the medial edge of the scapula. Taping will be performed after all initial measurements (T0) and will be renewed weekly (on days 0, 7, 14, 21). At the end of the 1st month, i.e. on day 28 (T1), the last measurements will be made with the patch and then the tape will be removed. One month after the end of the treatment, the patient will be called again (T2) and final measurements will be made without the tape.

Kyphosis Angle Measurement with Flexicurve:

At the beginning of the study,at the end of treatment (1st month) and 1 month after the end of treatment (2nd month).The Flexicurve ruler (Staedtler Mars Inc, Nurnberg, Germany),which is a plastic-coated bendable metal band approximately 60 cm long,will be used for the measurements.The ruler bends in only one direction and retains its shape when bent.The patient will stand as upright as possible and the spinous process of the seventh cervical vertebra(C7)and the upper part of the sacrum(S1)will be palpated and marked.The Flexicurve ruler will be placed along the C7-S1 vertebrae to form the shape of the spine,then the ruler will be placed flat on the paper and the lines transferred onto the paper.A vertical line will be drawn to connect the C7 and S1 landmarks.The intersection of this line with the spinal curve previously drawn with the flexicurve ruler will mark the transition between the thoracic and lumbar curves.A straight line drawn between C7 and the intersection point will be recorded as the thoracic kyphosis length (TL) in cm.Thoracic width (TW)will be recorded in cm as the length of the perpendicular line drawn from the apex of the kyphosis to TL.Kyphosis index will be calculated with the formula:(TL/TW) x 100.All measurements will be performed by two different specialists,repeated 2 times each and averaged.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-45
* Among the patients who applied to the physical medicine and rehabilitation outpatient clinic with poor posture or nonspecific back pain, the kyphosis angle was measured as ≥ 40 on the thoracic lateral radiograph
* Being literate
* Agreeing to participate in the research

Exclusion Criteria:

* Patients younger than 18 years and older than 45 years
* Spinal deformity, Scheuermann disease, disc herniation
* Previous spine surgery and trauma
* Neuromuscular, peripheral neuropathic disease
* Pregnant and postmenopausal women
* Vertigo disease (central or peripheral cause)
* Use of medication that may cause dizziness (in the last 3 months)
* Defect of vision
* Presence of physical deformity or additional disease that will prevent exercise
* Active skin disease in the area where tape will be applied

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Thoracic hyperkyphosis angle (Kyphosis Angle Measurement with Flexicurve) | 9 months
  They will be performed at the beginning of the study, at the end of treatment (1st month) and 1 month after the end of treatment (2nd month).
  Kyphosis index will be calculated with the formula: (TL/TW) x 100. Higher indices will indicate higher degrees of kyphosis.
  All measurements will be performed by two different specialists, repeated 2 times each and averaged.
  (How to measure is explained in detail in the 'detailed description' section).

SECONDARY OUTCOMES:
Static and Dynamic Balance Measurement with Biodex Device | 9 months
  Balance measurement of the patients will be performed with the Biodex Balance System SD (Biodex, Inc, Shirley, NY) (BBS). BBS is a movable circular platform that can move in antero-posterior and medio-lateral axes. In our study; bilateral stance static postural stability test (level 12, stable platform), bilateral stance dynamic postural stability test (level 4, unstable platform), single leg stance postural stability test (stable platform) and stability limit test will be measured. The postural stability measurement includes the overall stability index (OSI), anteroposterior stability index (APSI) and mediolateral stability index (MLSI). High values in these scores indicate poor balance. All balance tests will be performed with eyes open and barefoot and repeated 3 times with a 10-second rest interval.
Vas (Visual Analog Scale) Scoring | 9 months
  It will be evaluated before and at the end of treatment and at the end of the 2nd month and the patient will be asked to mark the degree of pain on a linear line with a value between 0-10.
Berg Balance Scale (Turkish) | 9 months
  The scale consists of 14 predetermined tasks, each task achievement is scored between 0-4, and will be performed 3 times: before treatment, at the end of the 1st month and at the end of the 2nd month.
SRS-22 (Turkish) | 9 months
  The SRS-22 questionnaire, which was developed by the Scoliosis Research Society (SRS) to be used in spinal curvatures and whose Turkish validity and reliability has been proven, will be filled out by patients before, at the end of treatment and at the 2nd month control.
International Physical Activity Questionnaire (Short) (IPAQ) | 9 months
  This questionnaire, the Turkish version of which has reliability and validity in assessing physical activity, will be completed by patients before, at the end and at 2 months of treatment to obtain information about their physical activity in daily life.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Marmara University Faculty of Medicine, Istanbul
  - Sultan 2.Abdülhamid Han Training and Research Hospital, Istanbul, Üsküdar

IPD SHARING:
Plan to Share IPD: No